CLINICAL TRIAL: NCT01429636
Title: Phase 3 Study of Applied Relaxation (AR) Technique That Treating Menopausal Symptoms
Brief Title: Applied Relaxation (AR) Technique Versus Its Modified Version for Treating Menopausal Symptoms
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Suprawita Saensak, Phase 3 Study of Applied Relaxation (AR) Technique versus Its Modified Version for Treating Menopausal Symptoms., Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARMR-Sympts
Record Dates: First submitted 2011-09-01; First posted 2011-09-07 (Estimated); Last update posted 2011-12-30 (Estimated); Status verified 2011-12

CONDITIONS: Hot Flashes; Night Sweats; Sleep Disturbances
Keywords: perimenopause; postmenopause; vasomotor symptoms; relaxation
MeSH Terms: conditions — Hot Flashes; Parasomnias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Applied Relaxation (AR) (Experimental)
  Interventions: Behavioral: Applied Relaxation (AR)
- Modified Relaxation (MR) (Experimental)
  Interventions: Behavioral: Modified Relaxation (MR)

INTERVENTIONS:
Behavioral: Modified Relaxation (MR) — The MR technique is modified from the AR technique that will require participants to attend only 1 session, lasting 60 minutes. After the training session, participants will be given a hand-out on MR. They will continue to practice MR at home once a day for 15-20 minutes during their leisure times, at least 5 days a week for the whole 12 weeks of the follow-up period.
  Other Names: Behavioral relaxation
  Arms: Modified Relaxation (MR)
Behavioral: Applied Relaxation (AR) — Participants will receive 12 sessions AR training. After that they will asked to practice at home once a day for 15-20 minutes during their leisure times, at least 5 days a week for the whole 12 weeks of the follow-up period.
  Other Names: Behavioral Applied Relaxation
  Arms: Applied Relaxation (AR)

SUMMARY:
The purpose of this study is to demonstrate better efficacy and effectiveness of modified applied relaxation technique over its original version for treating menopausal symptoms.

DETAILED DESCRIPTION:
Applied Relaxation (AR) is the most commonly used behavioral methods for treating menopausal symptoms. Many clinical trials reported that the technique effectively improved vasomotor and related symptoms. There is a strong evidence to support its continue use in clinical settings.

However, the original AR technique is too cumbersome. It involves intensive training once a week for 12 consecutive weeks. Each weekly session takes 60 minutes, and subjects are requested to do self-practice at home for at least 15-20 minutes/day. As such, >25% of recruited subjects drop out from the training course. The investigators have modified the original AR technique by reducing the duration of training to only once, lasting 60 minutes. Participants are requested to do self-practice at home for 15-20 minutes/day as in the original technique. Instead of coming to a weekly class, the investigators use telephone to communicate with the subjects once a week for 12 consecutive weeks. A preliminary study showed all 10 recruited subjects remained in the study (MR; modified relaxation technique) until completion. They all reported dramatic improvement in their vasomotor symptoms.

In this study, the investigators propose to compare our modified version of AR with the original method in a randomized controlled clinical trial. The subjects will be Thai menopausal women with vasomotor symptoms. The main outcomes are the reduction in the MRS score (intensity of hot flushes, night sweats and sleep disturbances) among those who remain in the program at the end of the study (efficacy evaluation). As nearly all patients will remain in the MR group, while >25% of those in the AR group will be expected to drop out from the study, the investigators should be able to demonstrate a superiority of MR over AR in terms of effectiveness as well.

ELIGIBILITY:
Inclusion Criteria:

* Perimenopausal women and postmenopausal women with either surgical or spontaneous menopause.
* Women who have at least 5 points of MRS score.

Exclusion Criteria:

* Women who are taking any hormone therapy for any reason in the past three months prior to entering the trails.
* Women with uncontrolled hypertension (>95mmHg diastolic pressure) or daily use of sedatives, tranquilizer or antidepressant medication.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Changes in global scores of Menopausal Rating Scale (MRS). | 12 weeks
  MRS measure after intervention at 1, 2 and 3 months for follow-up.

SECONDARY OUTCOMES:
Change in the frequency and severity of hot flushes. | 12 weeks
  Measure the frequency and severity of hot flushes after intervention at 1, 2 and 3 months.
Change in the frequency and severity of night sweats. | 12 weeks
  Measure the frequency and severity of night sweats after intervention at 1, 2, and 3 months.
Change in the frequency and severity of sleep disturbances. | 12 weeks
  Measure the frequency and severity of sleep disturbances after intervention at 1, 2, and 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Suprawita - Saensak, PhDcandidate, Principal Investigator — PhD in Clinical Epidemiology Program, Faculty of Medicine, Chiang Mai University (Thailand)
Locations (1):
- Mahassarakham Hospital, Maha Sarakham, Northeast, Thailand

REFERENCES:
- See also: NIH is the nation's medical research agency-supporting scientific studies that turn discovery into health. — http://www.nih.gov
- See also: PubMed comprises more than 21 million citations for biomedical literature from MEDLINE, life science journals, and online books. — http://www.ncbi.nlm.nih.gov/pubmed
- See also: Elsevier is committed to making genuine contributions to the science and health communities. — http://www.elsevier.com
- See also: The Journal of The North American Menopause Society is a peer-reviewed scientific journal owned by NAMS and published by Lippincott Williams & Wilkins (LWW). — http://www.menopause.org
- See also: The International Journal of Clinical and Health Psychology. — http://www.aepc.es/ijchp
- See also: The world's largest collection of STM books, journals, protocol and reference works. — http://www.springer.com/medicine/journal